CLINICAL TRIAL: NCT04540263
Title: Evaluation of Blood Cytokine Levels of Patients Who Underwent Sleeve Gastrectomy and Gastric Bypass Operations Due to Obesity
Brief Title: Cytokine Levels of Patients Who Underwent Obesity Surgery
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof. MD, Istanbul Training and Research Hospital
Other Study IDs: Obesity Cytokine
Record Dates: First submitted 2020-09-03; First posted 2020-09-07 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Obesity
Keywords: Sleeve Gastrectomy; Gastric bypass; Flow-cytometry; Cytokine
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sleeve Gastrectomy: Patients who underwent Sleeve gastrectomy operation
  Interventions: Diagnostic Test: Flow Cytometric analysis
- Gastric Bypass: Patients who underwent Gastric Bypass operation
  Interventions: Diagnostic Test: Flow Cytometric analysis

INTERVENTIONS:
Diagnostic Test: Flow Cytometric analysis — Measuring the level of IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1 (CCL2), IL-6, IL-8 (CXCL8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33 cytokines in the serum

SUMMARY:
Obesity is an important public health problem worldwide. There are large regional differences in the prevalence of overweight and obesity. Obesity is a growing problem in both developed and low-income countries. Obesity is a common condition characterized by excessive fat accumulation in adipose tissue. It is associated with metabolic, hematological and musculoskeletal complications, increased risk of dyslipidemia, heart disease, diabetes and some malignancies, leading to a shortened life span. Inflammation from adipose tissue has been identified as the main source of systemic inflammation and may also be associated with insulin resistance. Adipocytes and adipose tissue-related macrophages from obese individuals are an important source of inflammatory mediators such as TNF-α, IL-6, IL-1 and MCP-1. It has also been shown that decreased levels of IL-10, an anti-inflammatory cytokine, are associated with obesity and metabolic syndrome.We aimed to evaluate changes in 13 different proinflammatory and anti-inflammatory cytokines in patients who underwent sleeve gastrectomy or gastric bypass.

DETAILED DESCRIPTION:
Obesity is an important public health problem worldwide. There are large regional differences in the prevalence of overweight and obesity. Obesity is a growing problem in both developed and low-income countries. Obesity is a common condition characterized by excessive fat accumulation in adipose tissue. It is associated with metabolic, hematological and musculoskeletal complications, increased risk of dyslipidemia, heart disease, diabetes and some malignancies, leading to a shortened life span. Inflammation from adipose tissue has been identified as the main source of systemic inflammation and may also be associated with insulin resistance. Adipocytes and adipose tissue-related macrophages from obese individuals are an important source of inflammatory mediators such as TNF-α, IL-6, IL-1 and MCP-1. It has also been shown that decreased levels of IL-10, an anti-inflammatory cytokine, are associated with obesity and metabolic syndrome.There are many studies examining the changes in the weight and blood values of patients after bariatric surgery. Among these blood values, cytokines, which are inflammation mediators, were evaluated. However, in these studies, either sleeve gastrectomy or gastric bypass was evaluated separately and generally focused on TNF-α, IL-6, IL-1, IL10, and MCP-1 cytokines. There are conflicting results regarding the parameters examined in these studies. In some studies, no difference was found in the cytokines examined, while some regression was observed in proinflammatory cytokines. The situation is similar for IL10, which is one of the anti-inflammatory cytokines. An increase in IL10 values was observed in a study evaluating patients who underwent gastritic bypass, whereas no difference was found in a study evaluating sleeve gastrectomy patients.We aimed to evaluate changes in 13 different proinflammatory and anti-inflammatory cytokines before and 6 month after the surgery in patients who underwent sleeve gastrectomy or gastric bypass

ELIGIBILITY:
Inclusion Criteria:

* Patients who had sleeve gastrectomy or gastric bypass due to obesity

Exclusion Criteria:

* Cancer patients,
* Pregnant women,
* Have a history of immunodeficiency
* Patients with previous obesity surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had >35 body mass index and had obesity surgery (sleeve gastrectomy, gastric bypass) will be included
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Cytokine levels | 6 months
  Serum IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1 (CCL2), IL-6, IL-8 (CXCL8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33 levels

SECONDARY OUTCOMES:
Weight changes | 6 months
  The weight changes over time after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc.Prof., Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salman MA, Salman AA, Nafea MA, Sultan AAEA, Anwar HW, Ibrahim AH, Awad A, Ahmed RA, Seif El Nasr SM, Abouelregal TE, Shaaban HE, Mohamed FAH. Study of changes of obesity-related inflammatory cytokines after laparoscopic sleeve gastrectomy. ANZ J Surg. 2019 Oct;89(10):1265-1269. doi: 10.1111/ans.15427. Epub 2019 Sep 11. PMID 31508889
- [Background] Shimizu H, Hatao F, Imamura K, Takanishi K, Tsujino M. Early Effects of Sleeve Gastrectomy on Obesity-Related Cytokines and Bile Acid Metabolism in Morbidly Obese Japanese Patients. Obes Surg. 2017 Dec;27(12):3223-3229. doi: 10.1007/s11695-017-2756-9. PMID 28569359
- [Background] Cepeda-Lopez AC, Allende-Labastida J, Melse-Boonstra A, Osendarp SJ, Herter-Aeberli I, Moretti D, Rodriguez-Lastra R, Gonzalez-Salazar F, Villalpando S, Zimmermann MB. The effects of fat loss after bariatric surgery on inflammation, serum hepcidin, and iron absorption: a prospective 6-mo iron stable isotope study. Am J Clin Nutr. 2016 Oct;104(4):1030-1038. doi: 10.3945/ajcn.115.115592. Epub 2016 Aug 24. PMID 27557657